CLINICAL TRIAL: NCT05888545
Title: A Randomized Controlled Study on an Anti-adhesion Diaphragm in Preventing Intrauterine Adhesions
Brief Title: Clinical Study on a Novel Anti-adhesion Barrier Film
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K2023016
Record Dates: First submitted 2023-05-14; First posted 2023-06-05 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Intrauterine Adhesion
Keywords: Induced abortion; IUA; anti-adhesion barrier film
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-adhesion diaphragm (Experimental): Participants will be asked to place an anti-adhesion diaphragm in the uterus for 3-7 days after the abortion procedure.
  Interventions: Device: anti-adhesion diaphragm
- control group (No Intervention): Participants will be treated routinely with no other interventions.

INTERVENTIONS:
Device: anti-adhesion diaphragm — Participants will be asked to place an anti-adhesion diaphragm in the uterus for 3-7 days after the abortion procedure.
  Arms: anti-adhesion diaphragm

SUMMARY:
The aim of this clinical study was to verify the effectiveness and safety of the anti-adhesion diaphragm in preventing intrauterine adhesions.

DETAILED DESCRIPTION:
The main questions it aims to answer are

* The efficacy of the anti-adhesion diaphragm in preventing intrauterine adhesions;
* The duration of placement of the anti-adhesion septum in the uterus. Participants will be asked to place an anti-adhesion diaphragm in the uterus for 3-7 days after the abortion procedure. The control group will receive conventional treatment with no other interventions.

The researchers will compare the two groups to see if it is effective in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this trial and sign a written informed consent;
* Women aged 18 ≤ age ≤ 40 years;
* Those who had an abortion in early pregnancy, and those who had a cleanse.

Exclusion Criteria:

* Patients with scars;
* Patients with allergies;
* Patients with acute genitourinary tract infections;
* Patients with abnormalities of reproductive organs and abnormal uterine flexion after cesarean section;
* Patients with decreased menstrual flow after previous curettage;
* Patients with previous suspected or diagnosed uterine adhesions;
* Patients on immunosuppressive drugs;
* Patients with long-term use of antibiotics;
* Patients with malignant tumors of the reproductive organs;
* Patients with uterine adenomyosis, endometriosis, and uterine fibroids;
* Patients with severe systemic diseases;
* Patients with other conditions that are not suitable.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1176 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of uterine adhesions in the 3rd postoperative menstrual cycle. | one week before the third menstrual cycle post-index procedure
  The incidence of uterine adhesions was defined as the incidence of uterine adhesions in the control group of subjects with the uterine anti-adhesion septum placed to block the anterior and posterior uterine wall contact, and the incidence of adhesions in both groups was evaluated by ultrasound and/or hysteroscopy in the 3rd postoperative menstrual cycle.

SECONDARY OUTCOMES:
bleeding volume (Normal, decrease, increase) | two week, three months (third menstrual cycle) post-index procedure
  Menstruation
Postoperative Menstrual time（days） | two week, three months (third menstrual cycle) post-index procedure
  Postoperative Menstrual time（days）
Abdominal pain | two week, three months (third menstrual cycle) post-index procedure
  Abdominal pain due to postoperative menstruation
Physician satisfaction checklist | three months (third menstrual cycle) post-index procedure
  classified as very satisfied, satisfied, general and unsatisfied;
Patient acceptance chaecklist | three months (third menstrual cycle) post-index procedure
  willingness to use again and to recommend others;
Patient comfort after placement checklist | three months (third menstrual cycle) post-index procedure
  classified as comfortable, general, uncomfortable, and very uncomfortable.

OTHER OUTCOMES:
Number of Participants With Abnormal Laboratory Values | three months (third menstrual cycle) post-index procedure
  Abnormal Laboratory Values
body temperature ( ℃) | three months (third menstrual cycle) post-index procedure
  Vital signs
breathing (Times/minute) | three months (third menstrual cycle) post-index procedure
  Vital signs
blood pressure (mmHg) | three months (third menstrual cycle) post-index procedure
  Vital signs
heart rate ( Times/minute) | three months (third menstrual cycle) post-index procedure
  Vital signs
adverse reactions or adverse events | three months (third menstrual cycle) post-index procedure
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xu, PhD, Study Chair — The Fourth Affiliated Hospital Zhejiang University School of Medicine
Locations (8):
- China (8):
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - Lishui Hospital of TCM, Lishui, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang
  - The Second People's Hospital Of Quzhou, Zhejiang, Quzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang
  - Yuyao People's Hospital of Zhejiang Province, Yuyao, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hooker AB, de Leeuw RA, Twisk JWR, Brolmann HAM, Huirne JAF. Reproductive performance of women with and without intrauterine adhesions following recurrent dilatation and curettage for miscarriage: long-term follow-up of a randomized controlled trial. Hum Reprod. 2021 Jan 1;36(1):70-81. doi: 10.1093/humrep/deaa289. PMID 33320197
- [Background] Dreisler E, Kjer JJ. Asherman's syndrome: current perspectives on diagnosis and management. Int J Womens Health. 2019 Mar 20;11:191-198. doi: 10.2147/IJWH.S165474. eCollection 2019. PMID 30936754
- [Background] Lemmers M, Verschoor MA, Hooker AB, Opmeer BC, Limpens J, Huirne JA, Ankum WM, Mol BW. Dilatation and curettage increases the risk of subsequent preterm birth: a systematic review and meta-analysis. Hum Reprod. 2016 Jan;31(1):34-45. doi: 10.1093/humrep/dev274. Epub 2015 Nov 2. PMID 26534897